CLINICAL TRIAL: NCT05079217
Title: A Randomized, Double-Blinded Clinical Trial to Evaluate Additional Dose of Medium-dosage or High-dosage SARS-CoV-2 Inactivated Vaccine in Healthy Individuals Previously Vaccinated With CoronaVac
Brief Title: Safety and Immunogenicity Study of Booster Vaccination With Medium-dosage or High-dosage SARS-CoV-2 Inactivated Vaccine for Prevention of COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-4007
Record Dates: First submitted 2021-10-14; First posted 2021-10-15 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): 600 participants will receive one dose of booster vaccination with high-dosage inactivated SARS-CoV-2 vaccine .
  Interventions: Biological: High-dosage SARS-CoV-2 vaccine
- Control Group (Active Comparator): 600 participants will receive one dose of booster vaccination with medium-dosage inactivated SARS-CoV-2 vaccine .
  Interventions: Biological: Medium-dosage SARS-CoV-2 vaccine

INTERVENTIONS:
Biological: High-dosage SARS-CoV-2 vaccine — SARS-CoV-2 Inactivated Vaccine 1200SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Experimental Group
Biological: Medium-dosage SARS-CoV-2 vaccine — SARS-CoV-2 Inactivated Vaccine 600SU inactivated virus in 0.5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Control Group

SUMMARY:
This is a randomized, double-blinded, phase ⅠV clinical trial of SARS-CoV-2 inactivated vaccine manufactured by manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the safety and immunogenicity of booster vaccination with high-dosage SARS-CoV-2 vaccine in populations who have received two-dose Coronavac with 2nd dose vaccinated more than 6 month.

DETAILED DESCRIPTION:
This study a randomized, double-blinded, phase ⅠV clinical trial of SARS-CoV-2 inactivated vaccine .The purpose of this study is to evaluate the safety and immunogenicity of booster vaccination with high-dosage SARS-CoV-2 vaccine in populations who have received two-dose Coronavac with 2nd dose vaccinated more than 6 month.A total of 1200 subjects who have received two-dose Coronavac with 2nd dose vaccinated more than 6 month will be enrolled.All of subjects will be randomly divided into two groups in a 1:1 ratio .Subjects in experimental group will receive high-dosage SARS-CoV-2 inactivated vaccine.Subjects in control group will receive medium-dosage SARS-CoV-2 inactivated vaccine .

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-59;
* Proven legal identity;
* The subjects can understand and voluntarily sign the informed consent form and be willing to complete the study in accordance with the study plan;
* Have received two doses of inactivated SARS-CoV-2 vaccine(CoronaVac) manufactured by Sinovac Research & Development Co., Ltd at an interval of 21 to 35 days and is currently 6-8 months (180 to 240 days) after the second dose.

Exclusion Criteria:

* History of SARS-CoV-2 infection(laboratory confirmed);
* Have received three and more doses of inactivated SARS-CoV-2 vaccine;
* Severe adverse reactions, such as urticaria, dyspnea, and angioneurotic edema , occurred during the primary immunization;
* Autoimmune disease such as systemic lupus erythematosus or immunodeficiency / immunosuppression such as AIDS, post-transplant;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids(excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Acute diseases or acute exacerbation of chronic diseases within 7 days prior to booster vaccination;
* Axillary temperature >37.0°C;
* Already pregnant or are breastfeeding, planning to get pregnant within 1months (according to subjects' self-report and urine pregnancy test results);
* Participated in other clinical trials prior to enrollment and during the follow-up period, or planned to participate in other clinical trials during the clinical trial period;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity index-GMT of neutralizing antibodies（CZ02 strain） | Day 28 after booster vaccination
  GMT of neutralizing antibodies（CZ02 strain） 28 days after booster vaccination.

SECONDARY OUTCOMES:
Immunogenicity index-seropositive rate of neutralizing antibodies（CZ02 strain） | Day 28 after booster vaccination
  The seropositive rate of neutralizing antibodies（CZ02 strain） 28 days after booster vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies（CZ02 strain） | Day 28 after booster vaccination
  The seroconversion rate of neutralizing antibodies（CZ02 strain） 28 days after booster vaccination
Immunogenicity index-GMI of neutralizing antibodies（CZ02 strain） | Day 28 after booster vaccination
  GMI of neutralizing antibodies（CZ02 strain） 28 days after booster vaccination
Immunogenicity index-seropositive rate of neutralizing antibodies（Delta Strain） | Day 28 after booster vaccination
  The seropositive rate of neutralizing antibodies（Delta Strain） 28 days after booster vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies（Delta Strain） | Day 28 after booster vaccination
  The seroconversion rate of neutralizing antibodies（Delta Strain） 28 days after booster vaccination
Immunogenicity index-GMI of neutralizing antibodies（Delta Strain） | Day 28 after booster vaccination
  GMI of neutralizing antibodies（Delta Strain） 28 days after booster vaccination
Immunogenicity index-seroconversion rate of neutralizing antibodies（Omicron Strain） | Day 28 after booster vaccination
  The seroconversion rate of neutralizing antibodies（Omicron Strain） 28 days after booster vaccination
Immunogenicity index-seropositive rate of neutralizing antibodies（Omicron Strain） | Day 28 after booster vaccination
  The seropositive rate of neutralizing antibodies（Omicron Strain） 28 days after booster vaccination
Immunogenicity index-GMI of neutralizing antibodies（Omicron Strain） | Day 28 after booster vaccination
  GMI of neutralizing antibodies（Omicron Strain） 28 days after booster vaccination
Immunogenicity index-GMT of neutralizing antibodies（Omicron Strain） | Day 28 after booster vaccination
  GMT of neutralizing antibodies（Omicron Strain） 28 days after booster vaccination
Immunogenicity index-GMT of neutralizing antibodies（Delta Strain） | Day 28 after booster vaccination
  GMT of neutralizing antibodies（Delta Strain） 28 days after booster vaccination

OTHER OUTCOMES:
Immunogenicity index-the seropositive rate of neutralizing antibodies（CZ02 strain,Delta Strain and Omicron Strain） | 6 months after the booster vaccination
  The seroconversion rate of neutralizing antibodies（CZ02 strain,Delta Strain and Omicron Strain） 6 months after the booster vaccination
Immunogenicity index-GMT of neutralizing antibodies（CZ02 strain,Delta Strain and Omicron Strain） | 6 months after the booster vaccination
  GMI of neutralizing antibodies（CZ02 strain,Delta Strain and Omicron Strain） 6 months after the booster vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Master, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Xinqi City Center for Disease Control and Prevention, Xinqi, Jiangsu, China